CLINICAL TRIAL: NCT00645658
Title: Testosterone Replacement Therapy in Advanced Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Jonathan Myers, Principle Investigator, Palo Alto Veterans Institute for Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAB0015AGG/SGG; IRB# 10132
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Kidney Failure; Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — Testosterone

ARMS (2):
- Chronic kidney disease (Experimental): Patients with chronic kidney disease between the ages of 55 and 75 years.
  Interventions: Drug: Testim, 1% testosterone gel
- Control (No Intervention): Control participants with baseline data collection only (for baseline comparator).

INTERVENTIONS:
Drug: Testim, 1% testosterone gel — Subjects apply contents of gel packet (Testim, 1% testosterone gel) to skin daily.
  Arms: Chronic kidney disease

SUMMARY:
Muscle wasting is common in advanced chronic kidney disease (CKD) and adversely affects morbidity and mortality. In 2/3 of males with advanced CKD serum testosterone (TT) levels are reduced, and likely contributes to the wasting. As TT in relatively safe physiologic replacement doses, increases muscle mass in otherwise normal TT deficient subjects, we hypothesize that physiologic TT replacement will be effective in preventing and treating the loss of muscle mass and function in CKD patients, will improve quality of life and may reduce some cardiovascular disease (CVD) risk factors.

DETAILED DESCRIPTION:
All subjects will undergo baseline testing that will consist of functional capacity tests, blood tests and muscle biopsies (described in detail below). Subjects will then receive testosterone gel which will be applied daily to the skin of the abdomen or thighs every morning at the same time for 16 weeks. Two days after the hormone treatment is started, the blood testosterone (TT) level will be measured 6 hours after administration. Our goal will be the attainment of serum total TT levels in the mid- to upper normal young adult range. If the serum TT is not at goal, the dose of gel will be increased or decreased repeat testing will be performed within one week. All subjects will be tested for serum TT levels every 4 weeks to assure that the serum total TT remains at goal level. Measurements will be repeated at 8 and 16 weeks.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria: CKD subjects; males with calculated GFR (MRDR equation) between 15 and 40 ml/min/1.73m2 and stable or slowly progressive renal failure (decline in function of <1ml/min/month) including those patients requiring hemodialysis and serum testosterone levels of <300 ng/ml and capable of safely performing required exercise testing and serum testosterone levels of <300ng/ml and capable of safely performing required exercise testing.

Exclusion Criteria: Exclusion criteria: applicable to both CKD and control subjects. Any unstable chronic medical condition, previous kidney transplant. Uncontrolled diabetes mellitus, active vasculitis, active autoimmune disease, malignancy(<5 yrs), obesity (BMI > 35), alcoholism or other recreational drug use, active heart disease, angina, uncontrolled arrhythmias or myocardial infarct within past 3 months, peripheral vascular disease with claudication, active lung, liver or GI disease, sleep apnea, medically unstable subjects and subjects who received anabolic, catabolic or cytotoxic medications during the prior 3 months. History of prostate CA, PSA >4g/ml, or advanced BPH (AUA symptom score > 21) and abnormal prostate on digital rectal examination. Bone or joint abnormalities that would preclude exercise testing.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Rabkin, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Santa Clara Valley Medical Center, San Jose, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Kidney Disease: Patients with chronic kidney disease between the ages of 55 and 75 years.
  Testim (1% testosterone gel): Subjects apply contents of gel packet to skin daily.
Period: Overall Study
Arm/Group | Chronic Kidney Disease | Control
Started | 9 | 8
Completed | 8 | 6
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Did not complete all assesments | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Kidney Disease | Control | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.1) | 61.3 (8.9) | 60.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Black | 2 | 1 | 3
  Hispanic | 4 | 1 | 5
  White | 1 | 6 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Thigh Cross Sectional Area
Description: DEXA-determined thigh cross-sectional area
Time Frame: Baseline
Population: Outcome measure data were collected from CKD participants only; CKD participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: centimeters squared
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 8
centimeters squared | 58.2 (11)

2. Primary Outcome: Lean Body Mass
Description: DEXA-determined lean body mass
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 8
Kg | 48.2 (9)

3. Secondary Outcome: Fat Mass
Description: DEXA-determined total body fat mass
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 8
Kg | 21.2 (7.0)

4. Secondary Outcome: Quadriceps Strength
Description: Lower body strength (in lbs) using quadriceps leg extension.
Time Frame: Baseline
Reporting Status: Not Posted

5. Secondary Outcome: Kidney Disease-Specific Quality of Life
Description: Questionnaire - SF-36, which stands for the Short Form 36 Health Survey. It is a widely used standardized 36 item quality of life assessment. This particular measure focused on symptoms, and is scaled from zero to 100, with a higher score indicating better health functioning.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Kidney Disease
Number analyzed (Participants) | 8
units on a scale | 42.1 (8.1)

6. Secondary Outcome: Inflammatory Markers
Description: C-Reactive Protein (CRP). CRP is measured in mg/l and is a marker of inflammation. CRP generally ranges from <1.0 to 5 mg/L. A normal value is less than 2.0 mg/L.
Time Frame: pre treatment and monthly until end of treatment
Reporting Status: Not Posted

7. Secondary Outcome: Muscle Atrophy Signaling Pathways
Description: These include muscle growth regulatory factors, IGF-1 and myostatin, their receptors and components of the ubiquitin-proteasome and calpain proteolytic pathways and inflammatory cytokines.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 3-4 months
Description: Untoward or unfavorable medical occurrence in a participant
Arm/Group | Chronic Kidney Disease | Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

LIMITATIONS AND CAVEATS:
Limitation of funding period led to a small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes